CLINICAL TRIAL: NCT03907982
Title: Objective Randomised Blinded Investigation of Therapeutic Ablation Versus Cardioversion for Persistent Atrial Fibrillation
Brief Title: Investigation of Therapeutic Ablation Versus Cardioversion for AF
Acronym: ORBITA-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORBITA-AF Pilot study
Record Dates: First submitted 2019-03-22; First posted 2019-04-09 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Persistent Atrial Fibrillation; Cardiac Arrhythmia
Keywords: Cardiac ablation; Cardioversion; pacemaker; implantable cardioverter-defibrillator
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Internal Pilot as part of a future study, Randomised, blinded, controlled trial with 2 arms.
Who Masked: Participant, Investigator
Masking Description: Patient and physician - blinded randomisation to intervention (DCCV, or Pulmonary Vein Isolation plus DCCV)
  Once subject participation in the trial is complete, the patient and physician will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCCV + PVI (Experimental): DC cardioversion (DCCV) plus Pulmonary Vein Isolation (Cryoablation)
  At end of pulmonary vein isolation, DCCV performed (if patient still in AF). An implantable loop recorder will be inserted in the prepectoral area with local anaesthetic at the end of the procedure.
  Interventions: Procedure: DC Cardioversion; Procedure: Pulmonary vein isolation; Device: Implantable loop recorder
- DC cardioversion (DCCV) (Active Comparator): Acute treatment of heart rhythm by cardioversion. An implantable loop recorder will be inserted in the prepectoral area with local anaesthetic at the end of the procedure.
  Interventions: Procedure: DC Cardioversion; Device: Implantable loop recorder

INTERVENTIONS:
Procedure: DC Cardioversion — DC cardioversion (DCCV) is used to treat irregular heart rhythms (commonly atrial fibrillation). The procedure involves sedation or anaesthetic and placement of electrodes on the chest. An electrical impulse is passed across the electrodes to return the heart rhythm to normal.
Procedure: Pulmonary vein isolation — The cryoballoon (CE marked) is the key specified technique for performing pulmonary vein isolation in the ablation arm in this trial. This allows the physician electrophysiologist to perform a circumferential freeze around the pulmonary veins to electrically isolate the vein, thus preventing pulmonary vein ectopy from triggering AF.
  Arms: DCCV + PVI
Device: Implantable loop recorder — The Reveal device is inserted in the pre-pectoral position under the skin. This is performed with local anaesthetic and sedation at the end of the procedure clinic by the electrophysiologist performing the procedure. The device will provide a continuous recording of the heart rhythm and rate, and will be able to down load duration of AF episodes via a home monitoring system to establish the primary endpoint of the study.
  Other Names: LINQ

SUMMARY:
The main aim of the research is to investigate whether patients undergoing pulmonary vein isolation with cryoablation for atrial fibrillation (AF) will have lower rates of AF recurrence than those treated by DC cardioversion without an ablation procedure. The objectives of the Pilot Study are to validate the key study logistics with a view to optimising methods to be used in the main study.

DETAILED DESCRIPTION:
After adequate stroke prevention (e.g. anticoagulation) and rate control, the optimum strategy for patients who continue to be symptomatic with persistent AF has not been established. Cardioversion with antiarrhythmic medication is commonly used as a first-line rhythm control strategy despite very high recurrence rates of the index arrhythmia and high serious complications associated with this strategy. Further treatment options, such as catheter ablation or implantation of a pacemaker and ablation of the atrioventricular (AV) node, are considered once AF recurs. The benefits of first-line ablation in patients presenting with persistent AF has not been tested. We seek to perform a blinded, randomised trial comparing an electrical cardioversion-led strategy with a pulmonary-vein isolation strategy for the treatment of persistent atrial fibrillation.

No blinded randomised controlled trial comparing early-ablation strategies to cardioversion-led strategies has been performed. The rationale for blinding where possible in clinical trials is well established. The recently published ORBITA trial performed a blinded, multicentre randomised trial of percutaneous coronary intervention (PCI) in stable angina compared to a placebo procedure. This trial demonstrated that the efficacy of invasive procedures can be assessed with a placebo procedure and that this type of trial remains necessary. Knowledge of treatment assignment influences physician behaviour, drug recommendations and encourages bias in outcome reporting. The treatment effect size and the effects of confounding factors will be exaggerated and thus limit the interpretation of the true patient experienced outcomes either strategy. In a comparison of surgical procedures, a sham-control arm represents the gold standard of blinding. A systematic review of placebo-controlled surgical trials found no evidence of harm to participants assigned to the placebo group. For a procedure whose primary purpose is to give sustained symptomatic relief, definitive quantification of the true placebo-controlled effect size of AF ablation is necessary. There is a need to clarify the relationship between patient reported symptoms and the arrhythmia itself. Patient reported symptoms may not always be related to the severity of the arrhythmia or quality of life. No bias-resistant blinded, randomised, trial has yet been performed seeking to measure the benefits of AF ablation.

ELIGIBILITY:
Inclusion Criteria: Patients who meet the following inclusion criteria will be eligible for the study;

* Ability to give informed consent
* Age 18-80 years
* Persistent AF (atrial fibrillation lasting > 7days) of total continuous duration <2 years as documented in medical notes.
* Patients being considered for cardioversion.

Exclusion Criteria: Patients who meet the following exclusion criteria will be ineligible for study participation;

* Creatinine clearance (eGFR) < 30mls/min
* Contraindication or unable to take anticoagulation
* Known contraindication to or unable to tolerate amiodarone
* Uncontrolled hypertension
* Contraindication to catheter ablation
* BMI > 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schilling, FRCP MD, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust - St Bartholomew's Hospital and Whipps Cross Hospital, London, United Kingdom

REFERENCES:
- [Background] Wartolowska K, Judge A, Hopewell S, Collins GS, Dean BJ, Rombach I, Brindley D, Savulescu J, Beard DJ, Carr AJ. Use of placebo controls in the evaluation of surgery: systematic review. BMJ. 2014 May 21;348:g3253. doi: 10.1136/bmj.g3253. PMID 24850821
- [Background] Redberg RF. Sham controls in medical device trials. N Engl J Med. 2014 Sep 4;371(10):892-3. doi: 10.1056/NEJMp1406388. No abstract available. PMID 25184861
- [Background] Miller FG, Kaptchuk TJ. Sham procedures and the ethics of clinical trials. J R Soc Med. 2004 Dec;97(12):576-8. doi: 10.1177/014107680409701205. No abstract available. PMID 15574854
- [Background] Jones C, Pollit V, Fitzmaurice D, Cowan C; Guideline Development Group. The management of atrial fibrillation: summary of updated NICE guidance. BMJ. 2014 Jun 19;348:g3655. doi: 10.1136/bmj.g3655. No abstract available. PMID 24948694
- [Background] Brim RL, Miller FG. The potential benefit of the placebo effect in sham-controlled trials: implications for risk-benefit assessments and informed consent. J Med Ethics. 2013 Nov;39(11):703-7. doi: 10.1136/medethics-2012-101045. Epub 2012 Dec 13. PMID 23239742
- [Background] Al-Lamee R, Thompson D, Dehbi HM, Sen S, Tang K, Davies J, Keeble T, Mielewczik M, Kaprielian R, Malik IS, Nijjer SS, Petraco R, Cook C, Ahmad Y, Howard J, Baker C, Sharp A, Gerber R, Talwar S, Assomull R, Mayet J, Wensel R, Collier D, Shun-Shin M, Thom SA, Davies JE, Francis DP; ORBITA investigators. Percutaneous coronary intervention in stable angina (ORBITA): a double-blind, randomised controlled trial. Lancet. 2018 Jan 6;391(10115):31-40. doi: 10.1016/S0140-6736(17)32714-9. Epub 2017 Nov 2. PMID 29103656

RESULTS

PARTICIPANT FLOW:
Groups:
- DCCV + PVI: DC cardioversion (DCCV) plus Pulmonary Vein Isolation (Cryoablation)
  At end of pulmonary vein isolation, DCCV performed (if patient still in AF). An implantable loop recorder will be inserted in the prepectoral area with local anaesthetic at the end of the procedure.
  DC Cardioversion: DC cardioversion (DCCV) is used to treat irregular heart rhythms (commonly atrial fibrillation). The procedure involves sedation or anaesthetic and placement of electrodes on the chest. An electrical impulse is passed across the electrodes to return the heart rhythm to normal.
  Pulmonary vein isolation: The cryoballoon (CE marked) is the key specified technique for performing pulmonary vein isolation in the ablation arm in this trial. This allows the physician electrophysiologist to perform a circumferential freeze around the pulmonary veins to electrically isolate the vein, thus preventing pulmonary vein ectopy from triggering AF.
  Implantable loop recorder: The Reveal device is inserted in the pre-pectoral position under the skin. This is performed with local anaesthetic and sedation at the end of the procedure clinic by the electrophysiologist performing the procedure. The device will provide a continuous recording of the heart rhythm and rate, and will be able to down load duration of AF episodes via a home monitoring system to establish the primary endpoint of the study.
- DC Cardioversion (DCCV) + Placebo: Acute treatment of heart rhythm by cardioversion. An implantable loop recorder will be inserted in the prepectoral area with local anaesthetic at the end of the procedure.
  DC Cardioversion: DC cardioversion (DCCV) is used to treat irregular heart rhythms (commonly atrial fibrillation). The procedure involves sedation or anaesthetic and placement of electrodes on the chest. An electrical impulse is passed across the electrodes to return the heart rhythm to normal.
  Implantable loop recorder: The Reveal device is inserted in the pre-pectoral position under the skin. This is performed with local anaesthetic and sedation at the end of the procedure clinic by the electrophysiologist performing the procedure. The device will provide a continuous recording of the heart rhythm and rate, and will be able to down load duration of AF episodes via a home monitoring system to establish the primary endpoint of the study.
Period: Overall Study
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (6) | 72 (7) | 70.5 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of Persistent AF (of AF Episode Lasting > 7 Days).
Description: Data on epsiodes of Atrial Fibrillation (rate, duration) will be provided by the loop recorder, and downloaded via a home monitoring system
Time Frame: Within 12 months following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
Number analyzed (Participants) | 10 | 10
Participants | 3 | 6

2. Secondary Outcome: Death
Description: Death of the patient
Time Frame: Within 12 months of study recruitment
Measure: Count of Participants; unit: Participants
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

3. Secondary Outcome: Rates of Subject Hospital Re-admission
Description: Rates of admission of the subject back to hospital following the initial treatment for AF
Time Frame: Within 12 months following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
Number analyzed (Participants) | 10 | 10
Participants | 0 | 1

4. Secondary Outcome: Procedural Complications
Description: Assessment of rates of events that are considered procedural complications during the DCCV +/- Pulmonary Vein isolation (PVI) procedure
Time Frame: At the time of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
Number analyzed (Participants) | 10 | 10
Participants | 1 | 0

5. Secondary Outcome: Bleeding Events
Description: Rates of bleeding in subjects following the study DCCV +/- pulmonary vein isolation (PVI) procedures
Time Frame: Within 7 days of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
Number analyzed (Participants) | 10 | 10
Participants | 1 | 0

6. Secondary Outcome: Rates of Repeat Procedures
Description: Requirement for repeat procedures following the initial DCCV +/- pulmonary vein isolation (PVI) procedure for the study
Time Frame: within 12 months following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
Number analyzed (Participants) | 10 | 10
Participants | 4 | 7

7. Secondary Outcome: Clinical Success of Procedure
Description: Clinical procedural success as defined by 75% or greater reduction in the number of AF episodes as measured by the insertable cardiac monitoring system (LINQ) device.
Time Frame: Within 12 months following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
Number analyzed (Participants) | 10 | 10
Participants | 7 | 6

8. Secondary Outcome: Change in Quality of Life Measures (Using Short Form-12 Survey)
Description: Assessment of quality of life measures using Short Form Health Survey (SF12) questionnaire, which is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey (Ware, Kosinski, and Keller, 1996). The questions are combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. Scale range from 0 to 100, with higher scores indicating better quality of life.
Time Frame: Between baseline and 12 months after procedure
Population: A "low scale" indicates poorer health-related quality of life with Higher scores indicate a better outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | 12.21 (11.37) | 14.15 (2.73)

9. Secondary Outcome: Change in Quality of Life Measures (AF-PROMS)
Description: Assessment of Patient Reported Outcome Measures (PROMS) specific for Atrial Fibrillation (AF) in a series of 28 questions to assess the impact of AF on the subject's quality of life. Atrial Fibrillation Severity Scale (AFSS) uses a scale ranging from 0 to 35, where a higher score indicates more severe symptoms.
Time Frame: between baseline and 12 months after procedure
Population: A "low scale" indicates poorer health-related quality of life with higher scores indicate a better outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | -23 (22) | -2 (10)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | DCCV + PVI | DC Cardioversion (DCCV) + Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCCV + PVI (N=10) | DC Cardioversion (DCCV) + Placebo (N=10)
incisionla site bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — incisionla site bleeding at the ILR implant site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT03907982/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT03907982/SAP_001.pdf